CLINICAL TRIAL: NCT03810261
Title: Challenges in Achieving Adequate Vitamin D Status in the Adult Population - Part 2
Brief Title: Challenges in Achieving Adequate Vitamin D Status in the Adult Population/ Part 2
Acronym: VITAD/2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: VIST - Faculty of Applied Sciences (Other); Slovenian Research Agency (Other); Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VITAD-01-2018 Part 2
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oil-based vitamin D group (Experimental): Oil-based vitamin D, 1000 IU/day for 8 weeks
  Interventions: Dietary Supplement: Oil-based vitamin D
- Water-based vitamin D group (Experimental): Water-based vitamin D, 1000 IU/day for 8 weeks
  Interventions: Dietary Supplement: Water-based vitamin D
- Vitamin D capsules group (Experimental): Vitamin D capsules with starch-adsorbed vitamin D (powder), 1000 IU/day for 8 weeks
  Interventions: Dietary Supplement: Vitamin D capsules
- Control group (No Intervention): This group will receive no intervention.

INTERVENTIONS:
Dietary Supplement: Oil-based vitamin D — Participants will receive oil-based VALENS vitamin D, 1000 IU/day for 8 weeks.
  Arms: Oil-based vitamin D group
Dietary Supplement: Water-based vitamin D — Participants will receive water-based VALENS vitamin D, 1000 IU/day for 8 weeks.
  Arms: Water-based vitamin D group
Dietary Supplement: Vitamin D capsules — Participants will receive vitamin D capsules with starch-adsorbed vitamin D (powder), 1000 IU/day for 8 weeks.
  Arms: Vitamin D capsules group

SUMMARY:
The efficiency of different vitamin D formulations in treating suboptimal vitamin D status in adult population will be determined. It will provide insights into the influence of formulation on vitamin D absorption.

A randomised controlled intervention trial will be conducted on at least 72 subjects (18-65 years) with suboptimal Vitamin D status. Subjects will be selected from a pool of subjects in Part 1 of the study, after completion of winter sampling.

Study subjects will be randomised into four study groups (at least 18 subjects per study group). Three different treatments will be compared with a control group, which will not receive any supplemental Vitamin D. The three tested Vitamin D preparations in the treatment groups will be (A) oil-based VALENS vitamin D; (B) water-based VALENS vitamin D; and (C) Vitamin D capsules with starch-adsorbed vitamin D (powder). All these products are commercially available. Prior to study, actual level of vitamin D will be determined using appropriate analytical method. The treatment will be with 1000 IU Vitamin D per day, for two months, in all three groups. Second serum vitamin D level will be determined on last day of the treatment, and compared with pre-treatment vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* vitamin D suboptimal status
* Signed Informed consent form (ICF),
* Caucasian race
* Age between 18 and 65 years at the time of the signature of Informed consent form (ICF),
* Willingness to avoid a consumption of any food supplements containing Vitamin D during the study, except the ones prescribed by the study researchers, and to avoid use of solarium or other artificial UVB sources
* Willingness to follow all study procedures

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Known or suspected allergy to any ingredient of the tested products in Part 2,
* Pronounced avoidance of sunshine (eg reporting of allergy to the sun)
* Use of food supplements containing Vitamin D or fish oil or omega 3 fatty acids in last three months prior to inclusion,
* Special dietary habits used by a small part of the population (veganism, low-carb high-fat (LCHF) diet, caloric restriction diet, note: vegetarians are not excluded)
* Diets prescribed by the medical profession
* Disorders of the kidneys, thyroid, digestive tract, osteoporosis and other bone diseases, skin diseases
* Other diseases and conditions that affect the absorption and synthesis of vitamin D
* Exposure to stronger sunlight in the last three months prior to engaging in a survey (travel to countries with stronger sunshine, use of solarium),
* The consumption of margarine or plant substitutes for milk / milk products several times a day, as these foods are most often enriched with vitamin D,
* Visiting the solarium in the last three months before joining the survey,
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D serum concentration after 8 weeks of supplementation | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Principal Investigator — Researcher
Locations (1):
- Nutrition Institute, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No